CLINICAL TRIAL: NCT04319107
Title: Classifying Ectopia Lentis in Marfan Syndrome Into Five Grades of Increasing Severity
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: MARFAN_2020
Record Dates: First submitted 2020-03-20; First posted 2020-03-24 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Marfan Syndrome; Ectopia Lentis
MeSH Terms: conditions — Marfan Syndrome; Ectopia Lentis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Marfan Syndrome (MFS) patients: Patients who had a clinical diagnosis of MFS according to the revised Ghent criteria (ectopia lentis was not taken into account for the diagnosis), confirmed by FBN1 sequencing.
  Interventions: Other: ophthalmological examinations using a slit lamp bio microscopy and a three-mirror lens, standard procedure.
- Control patients: Relatives of MFS patients with none of the clinical features of MFS and in whom testing for the familial FBN1 mutation was negative.
  Interventions: Other: ophthalmological examinations using a slit lamp bio microscopy and a three-mirror lens, standard procedure.

INTERVENTIONS:
Other: ophthalmological examinations using a slit lamp bio microscopy and a three-mirror lens, standard procedure. — Pupillary dilatation was performed with instillation of tropicamide and phenylephrine. The ophthalmological examination included visual acuity measurement, using a slit lamp biomicroscopy to analyse the anterior segment and a three mirror lens to appreciate the quality of the dilation validated by the absence of pupillary reflex and to search for ectopia lentis. Ectopia Lentis grade is evaluated according to the 5-grade classification.

SUMMARY:
Marfan syndrome is characterized by musculoskeletal manifestations, cardiovascular disease and ocular abnormalities, particularly ectopia lentis. Diagnosis depends on clinical evaluation, family history and molecular data: mutation in the fibrillin-1 gene (FBN1). Ectopia lentis is the most common ocular manifestation in Marfan syndrome with FBN1 mutation and is relatively specific to this disease when associated with other features. However, clinical examinations for identifying ectopia lentis have not really been codified. The purpose of this study is to describe a 5-grade classification of increasing severity for ectopia lentis based on clinical examination and to evaluate the predictive value for the early grades of ectopia lentis in order to help characterize this major clinical diagnosis criterion.

ELIGIBILITY:
Inclusion Criteria:

* MFS patient, clinical diagnosis according to revised Ghent criteria, confirmed by FBN1 mutation.
* Relatives of MFS patients with none of the clinical features of MFS and in whom testing for the familial FBN1 mutation was negative.

Exclusion Criteria:

* Patients who had surgery for ectopia lentis
* Patients for whom dilation was not optimal.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: MFS patient or Relatives of MFS patients
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2013-12-31 (Actual)

PRIMARY OUTCOMES:
Ectopia lentis measurement | day 0
  Ectopia lentis measurement and classification into 5-stages. Evaluation of the predictive value of ectopia lentis, at early stages, in order to help characterize this major clinical diagnosis criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Audrey Putoux, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hopital Femme Mère Enfant, Bron, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zech JC, Putoux A, Decullier E, Fargeton AE, Edery P, Plauchu H, Dupuis-Girod S. Classifying Ectopia Lentis in Marfan Syndrome into Five Grades of Increasing Severity. J Clin Med. 2020 Mar 6;9(3):721. doi: 10.3390/jcm9030721. PMID 32155956